CLINICAL TRIAL: NCT05656794
Title: Consolidative Prostate Radiotherapy in Patients With Metastatic Prostate Cancer
Brief Title: Consolidative Prostate Radiotherapy in Metastatic Prostate Cancer
Acronym: CONSORT-PC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-5921
Record Dates: First submitted 2022-12-09; First posted 2022-12-19 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Prostate Metastases
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 - Investigational (Experimental): Radiation treatment (36 Gy in 6 fractions) to be delivered every other day over 2 weeks (excluding weekends).
  Interventions: Radiation: Radiotherapy
- Arm 2 - Standard (Other): Radiation treatment (36 Gy in 6 fractions) to be delivered once a week over 6 weeks.
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Standard of care radiotherapy administered as per institutional guidelines.

SUMMARY:
This is a prospective, randomized phase II trial investigating if radiation treatment delivered every other day for 2 weeks has the same side effects as radiation treatment delivered once weekly for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-proven metastatic prostate cancer
* Presence of low-volume or high-volume metastases (high volume defined as the presence of visceral metastases or ≥4 bone lesions with at least 1 lesion beyond the vertebral bodies and pelvis.)
* Planned to or receiving systemic treatment ADT +/- ARAT as per physician discretion (Previous chemotherapy allowed if completed more than 6 weeks prior to randomization.)
* Planned for EBRT
* ECOG 0 or 1
* Age 18 years or older

Exclusion Criteria:

* Prior radiotherapy to pelvis
* Active ulcerative colitis or Crohn's Disease, at discretion of treating physician
* Any condition where radiotherapy is contraindicated

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer excludes women
Enrollment: 40 (Estimated)
Dates: Start 2023-07-31 (Actual); Primary Completion 2031-08 (Estimated); Study Completion 2031-08 (Estimated)

PRIMARY OUTCOMES:
Rates of acute toxicity | 5 years
  Compare rates of acute toxicity between participants in Arm 1 and Arm 2. Acute toxicity will be measured using CTCAE V5.0

SECONDARY OUTCOMES:
Rates of late toxicity. | 5 years
  Compare rates of late toxicity between participants in Arm 1 and Arm 2. Acute toxicity will be measured using CTCAE V5.0
Measure failure-free survival | 5 years
  Compare failure-free survival, collected through medical records, for participants in Arm 1 and Arm 2

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Princess Margaret Hospital, Toronto, Ontario, Canada